CLINICAL TRIAL: NCT03892928
Title: Safety and Efficacy of Dexmedetomidine in Painless Colonoscopy: a Single-center, Randomized Study
Brief Title: Safety and Efficacy of Dexmedetomidine in Painless Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Clinical Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-12
Record Dates: First submitted 2019-02-20; First posted 2019-03-27 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine was infusion intravenously with a loading dose of 0.5 μg kg-1 for 10 min, then infusion at 0.3 μg kg-1 h-1 according to the ideal body weight of the patient until the end of colonoscopy. If Ramsay sedation scale score reached 3, colonoscope was inserted. During the whole process, maintenance Ramsay score of 3 to 4. Propofol 10 mg was administrated as the rescue dose if body movement occurred during colonoscopy.
  Interventions: Drug: Dexmedetomidine group
- Propofol group (Other): Propofol was administrated 1 mg kg-1 intravenously, then titrated given by 0.5 mg kg-1 until Ramsay score reached 3. During the whole process, propofol was given intermittently to maintain Ramsay score 3 to 4. If body movement happened, propofol 10mg was administrated every time.
  Interventions: Drug: Dexmedetomidine group

INTERVENTIONS:
Drug: Dexmedetomidine group — In the dexmedetomidine group, dexmedetomidine was infusion intravenously with a loading dose of 0.5 μg kg-1 for 10 min, then infusion at 0.3 μg kg-1 h-1 according to the ideal body weight of the patient until the end of colonoscopy. If Ramsay sedation scale score reached 3, colonoscope was inserted. During the whole process, maintenance Ramsay score of 3 to 4. Propofol 10 mg was administrated as the rescue dose if body movement occurred during colonoscopy. In the propofol group, propofol was administrated 1 mg kg-1 intravenously, then titrated given by 0.5 mg kg-1 until Ramsay score reached 3. During the whole process, propofol was given intermittently to maintain Ramsay score 3 to 4. If body movement happened, propofol 10mg was administrated every time.
  Other Names: Dexmedetomidine Hydrochloride group

SUMMARY:
104 patients who undergo painless colonoscopy from Decemenber 1,2019 to June 30,2022 will be randomized to two groups: propofol group and dexmedetomidine group.

In the dexmedetomidine group,dexmedetomidine was infusion intravenously with a loading dose of 0.5 μg kg-1 for 10 min, then infusion at 0.3 μg kg-1 h-1 according to the ideal body weight of the patient until the end of colonoscopy. In the propofol group, Propofol was administrated 1 mg kg-1 intravenously, then titrated given by 0.5 mg kg-1 during the whole process.

DETAILED DESCRIPTION:
104 patients who undergo painless colonoscopy from Decemenber 1,2019 to June 30,2022 will be randomized to two groups: propofol group and dexmedetomidine group.

In the dexmedetomidine group,dexmedetomidine was infusion intravenously with a loading dose of 0.5 μg kg-1 for 10 min, then infusion at 0.3 μg kg-1 h-1 according to the ideal body weight of the patient until the end of colonoscopy. In the propofol group, Propofol was administrated 1 mg kg-1 intravenously, then titrated given by 0.5 mg kg-1.For all patients, if Ramsay sedation scale score reached 3, colonoscope was inserted. During the whole process, maintenance Ramsay score of 3 to 4. Propofol 10 mg was administrated as the rescue dose if body movement occurred during colonoscopy

The primary outcome was the occurrence of hypotension. Secondary outcomes included the followings:(1) the duration and the maximum decreasing in BP. The time-weighted average which is measured by calculating the area under the threshold (AUT) divided by the total duration of colonoscopy. AUT = (depth of hypotension below a 20% decrease in systolic blood pressure or diastolic blood pressure from pre-procedure baseline or SBP of 90 mm Hg or DBP of 50 mm Hg× time in minutes spent of hypotension); (2) the incidence of bradycardia and hypoxemia, mask-assisted ventilation and body movement；(3) the discharge time , patients and endoscopists satisfaction score.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged above 18 years
2. American Society of Anesthesiologists (ASA) physical status of 1-2
3. Patients scheduled for sedation colonoscopy

Exclusion Criteria:

1. Emergency patients
2. Body weight < 40 kg or >100 kg
3. Allergy to dexmedetomidine, propofol in this trail, a previous adverse reaction to dexmedetomidine or propofol
4. Pregnancy or lactation
5. Drug abusers
6. Participation in other clinical studies within the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the occurrence of hypotension | The time during gastroscopy, an average of 12 minutes
  Hypotension is defined as a 20% decrease in systolic blood pressure or diastolic blood pressure from pre-procedure baseline, systolic blood pressure < 90 mmHg, and/or diastolic blood pressure < 50 mmHg

SECONDARY OUTCOMES:
The duration and the maximum decreasing in BP | The time during gastroscopy, an average of 12 minutes
  The time-weighted average which is measured by calculating the area under the threshold (AUT) divided by the total duration of colonoscopy. AUT = (depth of hypotension below a 20% decrease in systolic blood pressure or diastolic blood pressure from pre-procedure baseline or SBP of 90 mm Hg or DBP of 50 mm Hg× time in minutes spent of hypotension)
The incidence of bradycardia | The time during gastroscopy, an average of 12 minutes
  Bradycardia is defined as HR <50 beats/min
The incidence of hypoxemia | The time during gastroscopy, an average of 12 minutes
  Hypoxemia is defined as a decrease of SpO2 to <90%
The incidence of mask-assisted ventilation | The time during gastroscopy, an average of 12 minutes
  Mask ventilation is performed if the hypoxemia happened
The incidence of body movement | The time during gastroscopy, an average of 12 minutes
  Body movement is defined as the twisting of the patient's body due to the stimulation of the endoscopy, making it difficult to proceed with the procedure without additional propofol
The discharge time | From the end of colonoscopy to discharge，an average of 30 minutes
  The discharge time is calculated from the end of colonoscopy to discharge
Patients satisfaction score | When the patient is fully awake after colonoscopy，an average of 5 minutes
  Using an 11-point Likert scale, with 0 indicating "very dissatisfied" and 10 indicating "very satisfied"
Endoscopists satisfaction score | At the end of colonoscopy
  Using an 11-point Likert scale, with 0 indicating "very dissatisfied" and 10 indicating "very satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, Study Chair — China, Sichuan West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China